CLINICAL TRIAL: NCT04835038
Title: Effects of Sodium Bicarbonate Ringer's Injection and Sodium Lactated Ringer's Injection on Postoperative Acute Kidney Injury in Patients Undergoing Major Abdominal Surgery: a Randomized, Controlled, Open-label Clinical Study
Brief Title: Effects of BRS and LRS on Postoperative Acute Kidney Injury
Acronym: BRS/LRS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shiyong Li, Principal Investigator, Associate professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ChiCTR2100044465
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate Ringer's Injection group (Experimental): Intraoperative fluid therapy performed with BRS (Sodium Bicarbonate Ringer's Injection)
  Interventions: Drug: Sodium Bicarbonate Ringer's Injection
- Sodium Lactated Ringer's Injection group (Active Comparator): Intraoperative fluid therapy performed with LRS (Sodium Lactated Ringer's Injection)
  Interventions: Drug: Sodium Lactated Ringer's Injection

INTERVENTIONS:
Drug: Sodium Bicarbonate Ringer's Injection — Intraoperative fluid therapy performed with BRS (Sodium Bicarbonate Ringer's Injection)
  Arms: Sodium Bicarbonate Ringer's Injection group
Drug: Sodium Lactated Ringer's Injection — Intraoperative fluid therapy performed with LRS (Sodium Lactated Ringer's Injection)
  Arms: Sodium Lactated Ringer's Injection group

SUMMARY:
1. Title: Effects of Sodium Bicarbonate Ringer's Injection and Sodium Lactated Ringer's Injection on postoperative acute kidney injury in patients undergoing major abdominal surgery: a randomized, controlled, open-label clinical study
2. Objective: To evaluate the effect of BRS and LRS infusion on acute renal injury in patients undergoing major abdominal surgery
3. Primary outcome: Incidence of AKI at 28 days postoperative (defined as acute kidney injury, according to Kidgo 2012 definition and classification).
4. Study Design: Randomized, controlled, open-label clinical study.

DETAILED DESCRIPTION:
1. Subjects: patients who planned to undergo elective major abdominal surgery.
2. Study data collection period: Subjects signed the consent form until 28 days after discharge or died in hospital or withdrew from the study.
3. Number of research centers/sample size: 3400 patients were planned to be included.
4. Study process: Among patients undergoing elective surgery, the researchers will include patients who meet the inclusion criteria for elective major abdominal surgery and agree to participate in the study. The data to be collected in this study will be recorded by the researcher in the eCRF, including:

(1) Data to be collected during the screening period and preoperatively: patients' basic characteristics and demographic data (2) Data to be recorded during and/or after surgery: primary study indicators, secondary indicators, and other indicators.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade Ⅰ-Ⅲ.
2. patients aged between 20 and 70, signed informed consent form, and are willing to participate in the study.
3. BMI ≤ 30kg/m2.
4. elective major abdominal surgery for the first time (radical resection of ovarian cancer, radical resection of cervical cancer, radical resection of gastric cancer, radical resection of colorectal cancer, radical resection of bladder tumor and radical resection of prostate tumor).
5. NYHA cardiac function grade Ⅰ-Ⅲ.
6. the function of liver and kidney is normal before operation.
7. the blood coagulation function was normal before operation.
8. hemoglobin > 70g/L.
9. sinus rhythm was detected by electrocardiogram and there were no other malignant arrhythmias.

Exclusion Criteria:

1. Emergency surgery.
2. liver and kidney surgery.
3. complicated with chronic respiratory diseases and FEV1/FVC < 70%.
4. the operation time is less than 2 hours.
5. patients with mental illness or cognitive impairment.
6. uncontrolled hypertension with blood pressure higher than 180 × 100mmHg.
7. patients with hypothyroidism.
8. pregnant or lactating patients. -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute renal injury | 28 days after surgery
  The incidence of AKI at 28 days after surgery (Acute kidney injury is defined and graded according to KIDGO 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Shiyong Li, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No